CLINICAL TRIAL: NCT01657760
Title: Citalopram Effects on Craving and Dopamine Receptor Availability in Alcoholics
Acronym: CECDRAAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NURA-022-11F; 8331171 (Other Grant/Funding Number: VA HSR&D)
Record Dates: First submitted 2012-07-23; First posted 2012-08-06 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Dependence
Keywords: craving; dopamine; citalopram; ssri
MeSH Terms: conditions — Alcoholism | interventions — Citalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Intravenous saline control, in a double-blind, crossover study, with infusion days at least 2 weeks apart.
  Interventions: Drug: citalopram
- citalopram infusion (Active Comparator): 40 mg citalopram in 250 ml saline infused over 1 hour, in a double-blind, crossover study, with infusion days at least 2 weeks apart.
  Interventions: Drug: citalopram

INTERVENTIONS:
Drug: citalopram — citalopram, 40 mg IV, vs. saline control, each to be administered in a double-blinded, within-subjects design.

SUMMARY:
Alcohol use disorders (AUDs) are highly prevalent among U.S. civilians, and even more prevalent in the U.S. Veteran population. AUDs are frequently co-morbid with depressive symptoms in psychiatric clinical populations, resulting in an increased severity of both conditions. Indeed, returning Operation Enduring Freedom (OEF)/Operation Iraqi Freedom (OIF) Veterans have extraordinarily high rates of alcohol misuse and co-morbid psychiatric symptoms, indicating that future Veteran clinical populations will be particularly affected by AUDs. While FDA-approved medications are available to treat AUDs, their efficacy is low compared to available psychosocial treatments. Despite the lack of evidence for efficacy from controlled trials, antidepressants are frequently prescribed to clinical populations (including Veterans) with active AUDs. A better understanding of patient-level clinical variables that may confer poor response to treatment with antidepressants would allow clinicians better tools to distinguish those alcohol-dependent Veterans likely to do worse with antidepressant treatment.

DETAILED DESCRIPTION:
Description of Proposed Study A. Scientific Basis: Alcohol abuse and dependence represent a spectrum of maladaptive behaviors with enormous public health impact, especially for the U.S. Veteran population. Depressive symptoms are frequently comorbid with alcohol use disorders, but despite the frequent use of serotonin reuptake inhibitors (SSRIs) in clinical practice, clinical trials with these agents for alcohol use disorders have yielded mixed results concerning their impact on drinking behavior.

The characterization of alcohol-dependent subjects on the basis of demographic variables, severity of addiction, and psychiatric symptomatology has revealed a divergence in response to treatment with SSRIs among different subtypes of alcoholics (less severe "Type A" vs. more severe "Type B" alcohol dependence. Type A alcoholics have exhibited a trend toward decreased drinking behavior in clinical trials with SSRIs, whereas type B alcoholics showed a trend in the opposite direction. The literature does not offer an explanation for this divergence, and therefore, it is not clear how these research findings can be applied clinically.

As intravenous (iv) citalopram infusion (40 mg) bypasses hepatic metabolism, a single infusion produces a clinically relevant concentration in human brain, and the brain concentration remains stable for up to 4 h post-infusion, and is well-tolerated. A single infusion reduces striatal dopamine receptor binding potential by a magnitude comparable to the effect of chronic oral citalopram treatment, as measured by positron emission tomography (PET). The subjective experience of craving for alcohol in alcohol-dependent individuals has been associated with decreased dopamine receptor availability in the striatum via PET.

Significance of the research: Alcohol abuse and dependence occur at a higher rate in Veterans than in the overall U.S. population, and the presence of comorbid depressive symptoms amplifies the health risks to affected Veterans. While FDA-approved medications are available to treat alcohol dependence, their overall efficacy is low compared to available psychosocial treatments. Given that SSRIs are frequently utilized in Veteran populations with depressive symptoms and alcohol use disorders, there is the certainty that many Veterans with Type B alcohol dependence are receiving a pharmacological intervention that may exacerbate their drinking behavior, thereby increasing morbidity. A better understanding of patient-level clinical variables that may confer poor response to treatment with SSRIs would allow clinicians better tools to distinguish those alcohol-dependent Veterans likely to do worse, and prevent what was intended to be a beneficial medical intervention from worsening a Veteran's clinical course. This research is well-suited to a Veteran population because of the high proportion of Veterans with alcohol dependence.

C. Program Objectives: The nominee has a strong background in clinical addiction psychiatry, and he seeks to accomplish two objectives through the proposed training program: 1) to become an expert in the field of human alcohol addiction research, and 2) to learn techniques of PET research. The nominee's work environment at the West Los Angeles Veterans Administration Medical Center (WLAVA), in collaboration with colleagues at UCLA provides an ideal infrastructure for this training. He will be mentored by renowned experts in these areas, Drs. Arthur Brody, and Edythe London. The mentors have several NIH and VA grant-funded ongoing studies in alcohol and other addictive disorders research with strong ties to the VA PET research infrastructure. As part of training, the nominee will attend several courses and workshops at UCLA in foundational neuroimaging topics with relevance to PET (statistics, neuroimaging, neuroanatomy), as well as courses in the neurobiological bases of addiction. He will also attend annual conferences in Alcohol Dependence (Research Society on Alcoholism annual meeting) and neuroimaging (e.g., Society for Nuclear Medicine annual meeting), and meet with mentors regularly. The nominee plans to submit an NIH R01 and/or VA Merit Review grant toward the end of the award period. Long term, he plans to found an independent research career studying neuropharmacological approaches to treating and understanding substance use disorders, focusing primarily on alcohol.

D. Project Design and Methods: This project proposes to study 20 individuals in each of 3 groups (Type A alcohol dependence, Type B alcohol dependence, and healthy control subjects) for a double-blinded, placebo-controlled, within-subjects, outpatient study with iv citalopram (40 mg and saline, in counter-balanced order) and [18F]fallypride PET scanning. Participants should be in good physical health, have no history of complicated alcohol withdrawal symptoms (e.g., seizures, delirium tremens), be 21-55 years of age, and taking no psychoactive medications. Typology among alcohol-dependent subjects will be assessed after Kampman et al. (2007). The project aims: 1) To determine whether iv citalopram (40 mg) affects measures of craving for alcohol compared to a blinded saline iv control infusion; 2) to determine the change in striatal dopamine receptor D2/3 receptor availability (measured as binding potential for the radiotracer) with iv citalopram (40 mg) as compared to iv saline by [18F]fallypride PET scanning; and 3) to assess whether changes in striatal D2/3 receptor availability with iv citalopram (40 mg, compared to iv saline control) is related to measures of craving for alcohol among subjects.

E. Description of Intervention(s)/Treatment(s): Through Internet advertising, interested participants will be invited to call a phone number for anonymous phone screening, and individuals who pass phone screening will be invited to the WLAVA for a screening visit. Potential subjects will meet criteria for alcohol dependence (via SCID; except for control subjects), will have no current psychotropic medication use, will be in good physical health (as assessed by clinical history and physical examination and laboratory assay), and have no current dependence on other substances of abuse (SCID; aside from nicotine). After screening, qualified participants will be invited to participate in a structural magnetic resonance imaging (sMRI scan) for PET scan registration purposes, and two day-long experimental sessions at WLAVA, where they will undergo infusions with iv citalopram (40 mg and saline, double blinded); at least one week will separate infusion days to allow for participants to return to baseline functioning between sessions. After each infusion, participants will undergo ~30 min of paper- and computer-based questionnaires designed to assess measures of mood and other psychiatric symptoms, and ~15 min of assessment of both baseline and cue-induced craving for alcohol. Subsequently, participants will undergo [18F]fallypride PET scanning (~2h) to assess striatal D2/3 receptor availability. After completion of both infusions and PET scans, participants will be discharged from the study. Participants will be compensated for their participation according to VA research guidelines.

ELIGIBILITY:
Inclusion Criteria:

Must be U.S. Veteran

Alcohol Dependence:

* Age between 21 and 55;
* Meeting DSM-IV diagnostic criteria for alcohol dependence;
* Report drinking at least 48 standard drinks in a 30-day period, during the 90 days before enrollment, and
* Must have had at least 2 days of heavy drinking (at least 5 drinks/day for men, 4 drinks/day for women) in the last 30 days

Healthy Control:

* Age between 21 and 55;
* No Axis I DSM-IV diagnosis (except for nicotine dependence);
* Report drinking less than 10 drinks weekly over the past 90 days prior to study entry by Timeline Followback Method (TLFB).

Exclusion Criteria:

Exclusion criteria for Alcohol Dependence:

* Current treatment for alcohol problems or a history of treatment in the 30 days before enrollment or are treatment seeking;
* A current (last 12 months) DSM-IV diagnosis of dependence on any psychoactive substances other than alcohol and nicotine.

Exclusion criteria for Healthy Controls:

* Any history of treatment for alcohol or other substance use disorders;
* Any history of DSM-IV diagnosis of dependence on any psychoactive substances other than nicotine;
* Any history of DSM-IV diagnosis of Axis I mental illness.

Exclusion criteria for all subjects:

* A current (last 12 months) DSM-IV diagnosis of schizophrenia, bipolar disorder, other psychotic disorder, eating disorder, panic disorder with or without agoraphobia;
* Current use of psychoactive drugs, other than occasional marijuana use (< 3 uses per week), as determined by a positive urine screen for narcotics, amphetamines, or sedative hypnotics;
* Serious alcohol withdrawal symptoms as indicated by a score > 10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA);
* Clinically significant physical abnormalities as indicated by physical examination, hematological laboratory assay, or urinalysis, defined as: hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, alanine transaminase [ALT], aspartate aminotransferase [AST], and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal;
* A screening ECG that demonstrates anything other than normal sinus rhythm, normal conduction, and no clinically significant arrhythmias;
* History of epilepsy, seizures, or severe head trauma;
* History of alcohol intoxication delirium, alcohol withdrawal delirium or seizure, alcohol-induced persisting dementia, or alcohol-induced psychosis;
* Treatment with any of the following medications within the last 30 days prior to randomization: antidepressants, anti-convulsants, hypnotics, antipsychotics, psychomotor stimulants, or anti-anxiety agents;
* Previous treatment with citalopram discontinued due to an adverse event;
* Pregnancy, nursing, or refusal to use reliable barrier method of birth control, if female;
* Presence of metal fragments, pacemaker, or other ferromagnetic material which would prevent safe completion of an MRI scan;
* Recent history of radiation exposure which would make exposure to radiation from serial PET scans contraindicated;
* Non-zero breath-alcohol level on screening. We will exclude participants who present to study appointments intoxicated, as active alcohol intoxication may interact unpredictably with citalopram and produce unreliable results in assessments of mood or alcohol craving (e.g. Ray and Hutchison, 2007; Ray et al., 2011; see preliminary data C.2. above);
* Resting vital signs on any study visit outside of acceptable parameters: Pulse of 50-105 bpm, Blood pressures of 90-160 mm Hg systolic, 55-100 mm Hg diastolic;
* Any indication of suicidal ideation (i.e. as assessed by question 9 on the Beck Depression Inventory-II [BDI-II]), or elevated index of depressive symptoms, as evidenced by BDI-II score of 20;
* Presence in the body of a metal device (e.g., pacemaker, infusion pump, aneurysm clip, metal prosthesis or plate) that could either interfere with the acquisition of the MRI scan of the brain or for whom the MRI scan would pose a potential risk will be excluded.
* Radiation exposure: Participation in any other research study involving exposure to ionizing radiation in the past year if the total cumulative exposure from the past research studies and the current research study would exceed the limits described by the FDA in 21 CFR 361.1. Specifically, the total cumulative dose to the whole body, active blood-forming organs, lens of the eye, and gonads must remain below 5 rems, and the cumulated dose to all other organs must remain below 15 rems over the last year.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd S Zorick, MD PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zorick T, Okita K, Renard KB, Mandelkern MA, Brody AL, London ED. The Effects of Citalopram and Thalamic Dopamine D2/3 Receptor Availability on Decision-Making and Loss Aversion in Alcohol Dependence. Psychiatry J. 2022 Sep 20;2022:5663274. doi: 10.1155/2022/5663274. eCollection 2022. PMID 36249526

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Alcohol-dependent (AD) and healthy control (HC) participants were screened via the SCID-IV, excluding any participants with any Axis I psychiatric diagnosis within the last 6 months (aside from and alcohol dependence in the AD group). Fourteen potential AD and seventeen potential HC participants were enrolled and screened.
Pre-assignment Details: Enrolled participants who did not start study procedures either decided not to participate or failed screening.
Groups:
- Alcohol Dependent Citalopram First Placebo Second; Alcohol Dependent Placebo First Citalopram Second: DSM-IV alcohol dependent participants.
  Qualifying participants were invited back for three subsequent visits: a structural MRI scan, and two study medication/[18F]-fallypride PET scanning days (citalopram 40 mg iv, or saline placebo, double-blinded, administered in counter-balancing order) more than 1 week apart. All completing participants had breathalyzer-confirmed exhaled alcohol concentration of 0, and low alcohol withdrawal scores (confirming no intoxication and minimal alcohol withdrawal symptoms) on all study visits (see below). On study medication/PET scanning days, the following procedures were completed in order: 1. Breathalyzer, withdrawal, and psychiatric symptomatology screening; 2. Intravenous citalopram (or saline placebo) infusion (1 h). 3. Cue-induced craving assessment (~20 minutes). 4. [18F]-fallypride PET scanning (~3 h).
- Healthy Control Citalopram First Placebo Second; Healthy Control Placebo First Citalopram Second: participants with no Axis I mental illness or substance use disorder.
  Same procedures as AD group
Period: Overall Study
Arm/Group | Alcohol Dependent Citalopram First Placebo Second | Alcohol Dependent Placebo First Citalopram Second | Healthy Control Citalopram First Placebo Second | Healthy Control Placebo First Citalopram Second
Started | 5 | 7 | 7 | 7
Completed | 4 | 6 | 6 | 4
Not Completed | 1 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Patients with alcohol dependence and matched controls were enrolled
Groups:
- Alcohol Dependent: DSM-IV alcohol dependent
- Healthy Control: participants with no Axis I illness or substance use disorder
- Total: Total of all reporting groups
Arm/Group | Alcohol Dependent | Healthy Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 38 (7.6) | 41 (7.9) | 39.5 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 31 subjects enrolled, only 20 completed the study
  Participants
    Female | 2 | 5 | 7
    Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 31 enrolled, 20 completed the study
  Participants
    Race: White | 5 | 4 | 9
    Race: African American | 4 | 5 | 9
    Race: Asian | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Craving for Alcohol in Alcohol Dependence With Citalopram Compared to Placebo
Description: To assess whether craving for alcohol in alcohol dependence is affected by iv citalopram, compared to placebo.
  Cue-induced craving for alcohol was assessed using the Alcohol Urge Questionnaire, composed of 8 questions with responses on a 0 (none) to 7 (severe or highest level) which when scored provide an estimate of the level of craving for alcohol for the participant. A maximum score is thus 56, indicating the highest level of craving for alcohol, whereas the minimum score of 0 indicates no appreciable craving for alcohol.
Time Frame: 5 minutes after 1 hour of infusion intervention
Population: All participants completed both arms
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Alcohol Dependent Citalopram Infusion; Healthy Control Citalopram Infusion: 40 mg citalopram in 250 ml saline infused over 1 hour, in a double-blind, crossover study, with infusion days at least 2 weeks apart.
  citalopram: citalopram, 40 mg IV, vs. saline control, each to be administered in a double-blinded, within-subjects design.
- Alcohol Dependent Placebo; Healthy Control Placebo Infusion: Intravenous saline control, in a double-blind, crossover study, with infusion days at least 2 weeks apart.
  citalopram: citalopram, 40 mg IV, vs. saline control, each to be administered in a double-blinded, within-subjects design.
Arm/Group | Alcohol Dependent Citalopram Infusion | Alcohol Dependent Placebo | Healthy Control Citalopram Infusion | Healthy Control Placebo Infusion
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 21 (14.6) | 30.4 (17.9) | 10.8 (4.5) | 10.6 (3.7)

2. Secondary Outcome: Striatal Dopamine Receptor Availability in Alcohol Dependence With Citalopram, Compared to Placebo
Description: relative binding potential of dopamine D2/3 receptor specific tracer compared to cerebellum, where there is known to be almost no dopamine receptors.
Time Frame: 2-3 hours after 1 hour citalopram or placebo infusion
Measure: Mean (Standard Deviation); unit: striatal binding potential ratio
Groups:
- Alcohol Dependent Citalopram Infusion; Alcohol Dependent Placebo Infusion: DSM-IV alcohol dependent
- Healthy Control Citalopram Infusion; Healthy Control Placebo Infusion: participants with no Axis I illness or substance use disorder
Arm/Group | Alcohol Dependent Citalopram Infusion | Healthy Control Citalopram Infusion | Alcohol Dependent Placebo Infusion | Healthy Control Placebo Infusion
Number analyzed (Participants) | 10 | 10 | 10 | 10
striatal binding potential ratio | 22.4 (4.0) | 25.7 (5.1) | 22.5 (3.8) | 21.3 (4.7)
Statistical Analysis 1: Comparison: Alcohol Dependent Citalopram Infusion vs Healthy Control Citalopram Infusion; Test type: Equivalence — 80% power to detect difference p<0.05 two tailed; p = 0.87, ANOVA — ANOVA, uncorrected for MC; Mean Difference (Final Values) = 0.01, Standard Deviation 0.03

ADVERSE EVENTS:
Time Frame: two weeks of study procedures per participant
Description: Adverse events were collected on all study days, both upon initial participant contact, during the study procedures, and upon completing each day's study procedures.
Arm/Group | Placebo | Citalopram Infusion
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 7/20 | 12/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=20) | Citalopram Infusion (N=20)
nausea (Gastrointestinal disorders) | 1 (1) | 8 (8) — subjective experience of nausea
anxiety (Nervous system disorders) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 2 (2) | 5 (5) — temporary dizziness
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) — stomach upset
fatigue (Nervous system disorders) | 2 (2) | 7 (7)
muscle tension (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
insomnia (Nervous system disorders) | 0 (0) | 1 (1) — occurring after study medication given

LIMITATIONS AND CAVEATS:
A limitation of the study is the modest sample size. Due to the collinearity between smoking and alcohol dependence in the sample, we are also unable to effectively disentangle any specific effect of smoking status on any of the measures reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT01657760/Prot_SAP_000.pdf